CLINICAL TRIAL: NCT05231252
Title: The Effect of Direct Cyclophotocoagulation Using Endolaser in Silicon Induced Glaucoma: a Pilot Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Ahmed Hashiem, Lecturer of ophthalmology,Principal Investigator ,Ophthalmology consultant., Kafrelsheikh University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 27-12-22
Record Dates: First submitted 2022-01-28; First posted 2022-02-09 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Intervention Model Description: pilot
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Cyclophotocoagulation — Transcleral cyclophotocoagulation is used to treat glaucoma secondary to silicone oil.

SUMMARY:
Transcleral cyclophotocoagulation has been used to treat glaucoma secondary to silicone oil

ELIGIBILITY:
Inclusion Criteria:

. Patients above 18 years of age. .Silicon filled for more than 2 months. .IOP more than 21 mmHg on triple topical antiglaucoma eye drops.

Exclusion Criteria: . History of glaucoma prior to the initial retinal surgery. . Immediate rise of IOP after SOI. . History of previous laser application to the ciliary body. . Any contraindications for silicone oil removal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
IOP lowering in patients with silicon induced glaucoma | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A.Mohamed, PhD, Study Director — Ain Shams University,Faculty of medicine
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
will not be shared til manuscript publishment